CLINICAL TRIAL: NCT03335423
Title: Inter- and Intra-individual Variations in Metformin Pharmacokinetics - The Importance of Genes and Drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ida Kuhlmann, Principal investigator, University of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1779
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2018-01

CONDITIONS: Metformin; Organic Cation Transporter 1; Codeine
MeSH Terms: interventions — Metformin; Codeine

STUDY DESIGN:
Intervention Model Description: In part 1 a single group of healthy volunteers will ingest a single dosis of metformin and then have a blood sample drawn after 3 and 10 hours.
  In part 3, 18 healthy subjects will be randomized to ingest: a) oral metformin b) intravenous metformin c) 4 pills of codeine with the 5th taken together with oral metformin and d) 4 pills of codeine with the 5th taken together with intravenous metformin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral Metformin (Experimental): Oral metformin 1000mg will be given as a single dosis
  Interventions: Drug: Oral metformin
- Intravenous metformin (Experimental): Intravenous metformin 500mg will be injected as a single dosis
  Interventions: Drug: Intravenous metformin
- Oral codeine and oral metformin (Experimental): Codeine 25 mg will be given at 5 occasions with approximately 6 hours between each dosing. The fifth and last dose will be given together with 1000 mg oral metformin
  Interventions: Drug: Oral codeine and oral metformin
- Oral codeine and intravenous metformin (Experimental): Codeine 25 mg will be given at 5 occasions with approximately 6 hours between each dosing. The fifth and last dose will be given together with 500 mg metformin administrated as an injection.
  Interventions: Drug: Oral codeine and intravenous metformin

INTERVENTIONS:
Drug: Oral metformin — The study was designed as a randomized, cross-over trial with a washout period of at least 1 week between the phases. Metformin was given both orally and through an intravenous route to be able to determine the absolute bioavailability of metformin. Metformin was given alone and together with codeine to investigate a potential interaction between the drugs. Lactate was measured as a proxy for metformin effect on the intestinal mucosa, both after oral and intravenous metformin
  Arms: Oral Metformin
Drug: Intravenous metformin — The study was designed as a randomized, cross-over trial with a washout period of at least 1 week between the phases. Metformin was given both orally and through an intravenous route to be able to determine the absolute bioavailability of metformin. Metformin was given alone and together with codeine to investigate a potential interaction between the drugs. Lactate was measured as a proxy for metformin effect on the intestinal mucosa, both after oral and intravenous metformin
  Arms: Intravenous metformin
Drug: Oral codeine and oral metformin — The study was designed as a randomized, cross-over trial with a washout period of at least 1 week between the phases. Metformin was given both orally and through an intravenous route to be able to determine the absolute bioavailability of metformin. Metformin was given alone and together with codeine to investigate a potential interaction between the drugs. Lactate was measured as a proxy for metformin effect on the intestinal mucosa, both after oral and intravenous metformin
  Arms: Oral codeine and oral metformin
Drug: Oral codeine and intravenous metformin — The study was designed as a randomized, cross-over trial with a washout period of at least 1 week between the phases. Metformin was given both orally and through an intravenous route to be able to determine the absolute bioavailability of metformin. Metformin was given alone and together with codeine to investigate a potential interaction between the drugs. Lactate was measured as a proxy for metformin effect on the intestinal mucosa, both after oral and intravenous metformin
  Arms: Oral codeine and intravenous metformin

SUMMARY:
The investigators aim to investigate the interindividual variation in metformin AUC in a large cohort of healthy volunteers after a single dose of metformin. Part 1 is driven by the hypothesis that metformin AUC and renal clearance exhibit significant interindividual variation. However this has never been documented in a large cohort of healthy volunteers.

The investigators aim to investigate the potential interaction between codeine and metformin in the intestine. The hypothesis underlying part 3 is that the increased risk of early discontinuation of metformin during co-administration with codeine is primarily due to local inhibition of OCT1 via codeine at the intestinal level.

DETAILED DESCRIPTION:
Part 1: The investigators intend to investigate the inter-individual variation in metformin Area Under Plasma Concentration Curve (AUC) following a single dose of oral metformin based on the plasma concentration of metformin after 3 and 10 hours and urine collection for 24 hours . Part 2: The investigators intend to contribute with DNA and metformin AUC determinations from subjects from part 1 to a major international study that aime to highlight the Genome Wide Association (GWA) between the entire genome and variations in metformin pharmacokinetics (AUC) in a large group of healthy subjects and patients. Part 3: The investigators aim to investigate the potential interaction between codeine and metformin in the intestine.

The investigators secondary objective in part 3 is to investigate if the plasma concentration of morphine increases when codeine and metformin are given together due to competitive inhibition of the Organic cation transporter 1 (OCT1) transport protein (in the liver). Furthermore, the investigators will measure lactate after metformin ingestion as a proxy for metformin's effect on the intestinal mucosa, both after oral and intravenous metformin

ELIGIBILITY:
Inclusion Criteria Part 1 (and 2): Men and women. Apparent good general health. eGFR, creatinine, Hba1c, must be within the reference range or clinically insignificantly differ from this. Written consent must be given. Age 18-65. BMI 18,5 - 29,9kg/m².

-

Exclusion Criteria part 1 (and 2): Daily consumption of medicine (prescription, over the counter and herbal medicines, dietary supplements (oral contraceptives and regular vitamin pills are accepted)). Alcohol abuse. Hypersensitivity for metformin. For women: positive pregnancy test and not using safe contraceptives for 24 hours after intake of metformin and breastfeeding.

Inclusion Criteria Part 3:Apparent good general health. eGFR, creatinine, Hba1c, glucose, ALAT and bilirubin must be within the reference range or clinically insignificantly differ from this. Written consent must be given. Age 18-30 . BMI 18,5 - 29,9kg/m².

Exclusion Criteria part 3: Daily consumption of medicine (prescription, over the counter and herbal medicines, dietary supplements (regular vitamin pills are accepted)). Alcohol abuse. Hypersensitivity for metformin, codeine or morphine. Genetically proven CYP2D6 slow or ultra-fast metabolizers. Genetically proven loss-of-function allele in OCT1

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
Metformin AUC | blood samples will be collected after 3 and 10 hours for each subject (N=300) after oral metformin ingestion. Urine is collected for 24 hours.
  Outcomes of part 1: Variation in metformin AUC in a large cohort of healthy volunteers after a single dose of metformin
Metformin AUC | Blood samples will be drawn in each of the 4 arms from ingestion of the drug/drugs and for 24 hours at suitable times. Urine is collected after ingestion of metformin for 24 hours.
  Outcome of part 3; differences in AUC for metformin when given alone and together with codeine

SECONDARY OUTCOMES:
Codeine AUC | Blood samples are collected for 6 hours after ingestion of the first codeine pill. Blood samples are also collected and measured for codeine, morphing, M3G,M6G for 6 hours after both oral and intravenous metformin
  secondary outcome of part 3: differences in codeine AUC when codeine is given alone and together with metformin
Lactate AUC | Blood samples for lactate will be drawn in each arm after metformin ingestion for 24 hours at suitable times
  Secondary outcome of part 3: differences in lactate AUC after metformin is given orally and intravenously

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brøsen, professor, chief physcian, Study Chair — University of Southern Denmark
Locations (1):
- The department of clinical pharmacy and pharmacology, Odense, Denmark